CLINICAL TRIAL: NCT05488847
Title: Multimodal Nonopioid Pain Protocol Following Shoulder Arthroplasty Surgery
Brief Title: Opioid-Free Pain Protocol After Shoulder Arthroplasty
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Stephanie Muh, MD, Deputy Chief, Department of Orthopaedics Surgery Service, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15592
Record Dates: First submitted 2022-07-20; First posted 2022-08-05 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Shoulder Arthropathy; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Celecoxib; Pregabalin; Tramadol; Dexamethasone; Calcium Dobesilate; Acetaminophen; Ropivacaine; Epinephrine; Ketorolac; tizanidine; Magnesium; Magnesium Oxide; Ibuprofen; Oxycodone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Multimodal, Non-Narcotic (Experimental): This group will be given the preoperative, intraoperative, and discharge meds described below. This group will NOT receive any opioid-containing meds. Preoperative meds: Celecoxib: 400 mg by mouth, Pregabalin: 75 mg by mouth, Tramadol: 50 mg by mouth. Intraoperative meds: Dexamethasone: 10 mg IV, Acetaminophen: 1,000 mg IV, Ropivacaine 5 mg/mL (0.5%): 300 mg local infiltration, Epinephrine 1 mg/mL (1:1000): 1 mg local infiltration, Ketorolac 30 mg/mL: 30 mg local infiltration. Discharge meds: Dexamethasone: 4 mg by mouth twice per day for 4 days (for same day discharge only), 10 mg IV on postoperative day 1 (for overnight patients only), Pregabalin: 75 mg by mouth twice per day for 14 days, Tizanidine: 2 mg by mouth every 6 hours for 14 days, Magnesium: 200 mg by mouth twice per day for 14 days, Ibuprofen: 600 mg by mouth every 6 hours not to exceed 3200 mg per day for 1 month, Acetaminophen: 975 mg by mouth every 8 hours not to exceed 3000 mg per day for 1 month.
  Interventions: Drug: Celecoxib; Drug: Pregabalin; Drug: Tramadol; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Ropivicaine; Drug: Epinephrine; Drug: Ketorolac; Drug: Tizanidine; Drug: Magnesium; Drug: Ibuprofen
- Multimodal Plus Narcotic (Active Comparator): This group will be given the preop, intraop, and discharge meds described below. They will also be given 35 pills of oxycodone hydrochloride 5mg to be taken every 6 hours as needed at discharge. Preoperative: Celecoxib: 400 mg PO, Pregabalin: 75 mg PO, Tramadol: 50 mg PO. Intraoperative: Dexamethasone: 10 mg IV, Acetaminophen: 1,000 mg IV, Ropivacaine 5 mg/mL (0.5%): 300 mg local infiltration, Epinephrine 1 mg/mL (1:1000): 1 mg local infiltration, Ketorolac 30 mg/mL: 30 mg local infiltration. Discharge: Dexamethasone: 4 mg PO twice per day for 4 days (for same day discharge only), 10 mg IV on postop day 1 (for overnight patients only), Pregabalin: 75 mg PO twice per day for 14 days, Tizanidine: 2 mg PO every 6 hours for 14 days, Magnesium: 200 mg PO twice per day for 14 days, Ibuprofen: 600 mg PO every 6 hours not to exceed 3200 mg per day for 1 month, Acetaminophen: 975 mg PO every 8 hours not to exceed 3000 mg per day for 1 month.
  Interventions: Drug: Celecoxib; Drug: Pregabalin; Drug: Tramadol; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Ropivicaine; Drug: Epinephrine; Drug: Ketorolac; Drug: Tizanidine; Drug: Magnesium; Drug: Ibuprofen; Drug: Oxycodone Hydrochloride 5 Mg

INTERVENTIONS:
Drug: Celecoxib — preoperative pain medication given to all patients
  Other Names: Celebrex
Drug: Pregabalin — preoperative and discharge pain medication given to all patients
  Other Names: Lyrica
Drug: Tramadol — preoperative pain medication given to all patients
  Other Names: Ultram
Drug: Dexamethasone — Intraoperative and discharge pain medication given to all patients
  Other Names: Decadron
Drug: Acetaminophen — Intraoperative and discharge pain medication given to all patients
  Other Names: tylenol
Drug: Ropivicaine — Intraoperative pain medication given to all patients
  Other Names: naropin
Drug: Epinephrine — Intraoperative pain medication given to all patients
Drug: Ketorolac — Intraoperative pain medication given to all patients
Drug: Tizanidine — Discharge pain medication given to all patients
  Other Names: Zanaflex
Drug: Magnesium — Discharge pain medication given to all patients
  Other Names: magnesium oxide
Drug: Ibuprofen — Discharge pain medication given to all patients
  Other Names: Motrin
Drug: Oxycodone Hydrochloride 5 Mg — Only given to active comparator group
  Other Names: Roxicodone
  Arms: Multimodal Plus Narcotic

SUMMARY:
This randomized, single blinded, clinical trial aims to investigate the efficacy of a multimodal pain control regimen for shoulder arthroplasty. Patients who receive a multimodal pain control regimen alone (study group) will be compared to patients who receive a multimodal pain control regimen plus a standard prescription of an opioid containing medication (comparison group). The primary outcome is average daily Numerical Rating Scale (NRS) pain score in the first 10 days after surgery. We hypothesize that there will be no significant difference in the primary outcome between the two groups.

DETAILED DESCRIPTION:
The United States is in the midst of an ongoing opioid crisis. In 2019, approximately 153 million opioid prescriptions were dispensed (46.7 per 100 persons) and 50,000 people died from opioid-involved overdoses. Orthopaedic and spine conditions account for 27.7% of opioid prescriptions and prior studies demonstrate that musculoskeletal pain is frequently reported by opioid abusers as their initial reason for consuming opioids. For these reasons, orthopaedic surgeons are uniquely posed to combat this crisis. Multimodal pain control is a strategy that utilizes multiple pain medications to provide analgesia. The theory behind this strategy is that agents with different mechanisms of action work synergistically to reduce pain by blocking multiple pain pathways. Several randomized controlled trials have investigated the efficacy of multimodal pain control for orthopaedic procedures, including anterior cruciate ligament reconstruction, labral repair, meniscus repair, and rotator cuff repair. In these studies, patients who received a multimodal nonopioid regimen had equivalent or better postoperative pain control compared to a standard opioid regimen. Furthermore, no severe side effects were reported in patients who received the multimodal nonopioid regimen. This randomized, single blinded, standard of care-controlled clinical trial aims to investigate the efficacy of a multimodal pain control (similar to the regimen utilized in the aforementioned studies) for controlling pain following shoulder arthroplasty. Adult patients indicated for anatomic or reverse total shoulder arthroplasty will be randomized to either the experimental or comparison group. The experimental group will receive a multimodal, non-narcotic pain control regimen consisting of Celecoxib, Pregabalin, and Tramadol preoperatively; Dexamethasone, Acetaminophen, Ropivacaine, Epinephrine, and Ketorolac intraoperatively; and Dexamethasone, Pregabalin, Tizanidine, Magnesium, Ibuprofen, and Acetaminophen postoperatively. In addition to the aforementioned multimodal pain control regimen, the comparison group will receive a standard prescription of Oxycodone to be taken as needed postoperatively. If patients in the experimental group feel their pain is uncontrolled, they have the option of calling in to request a prescription of Oxycodone. Pain, pain medication use, and medication side effects will be closely monitored for the first 10 days after surgery by having patients respond to daily automated text messages. Additionally, all study participants will complete patient-reported outcome measures (PROMs) surveys and undergo physical examination of their shoulder during routine clinic visits preoperatively and at 1 week, 6 weeks, 3 months, 6 months, 1 year, and 2 years postoperatively. The primary outcome of this study is postoperative pain scores on the Numerical Rating Scale (NRS) for the first 10 days postoperatively. We hypothesize that there will be no significant difference between the groups with regard to the primary outcome. Secondary outcomes measured during the first 10 days postoperative include morphine milligram equivalents (MMEs) of opioids consumed, Patient-Reported Outcome Measurement Information System Pain Interference (PROMIS-PI) score at first postoperative clinic visit (7-10 days postoperatively), duration of patient reported adverse events (ie, constipation, nausea, diarrhea, upset stomach, drowsiness, loopiness), perioperative complications, and satisfaction with pain control. Secondary outcomes measured at routine postoperative clinic visits out to 2 years after surgery include postoperative complications, need for revision surgery, PROM scores (ie, PROMIS upper extremity, PROMIS PI, PROMIS D, American Shoulder and Elbow Surgeons Shoulder Score, Shoulder Arthroplasty Smart, Constant-Murley), hospital and emergency department readmission (30-day, 60-day, 90-day), duration of narcotic pain medication use shoulder strength, and shoulder range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Consented and scheduled for primary anatomic or reverse total shoulder arthroplasty at a Henry Ford hospital location

Exclusion Criteria:

* Unable to receive or reply to mobile phone text messages.
* Unable to read or speak English
* Medical history of known allergies or intolerance to any of the medications prescribed as a part of this study (ie, Percocet, Ibuprofen, Pregabalin, Dexamethasone, Acetaminophen, Tizanidine, Magnesium, Celecoxib, Tramadol, Ropivacaine, Epinephrine, Ketorolac)
* Substantial alcohol or drug abuse
* Recent or current pregnancy
* History of narcotic use within 3 months prior to surgery
* Renal or hepatic impairment or dysfunction
* Use of blood thinner medication
* Peptic ulcer disease
* Gastrointestinal bleeding
* History of gastric bypass surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2026-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J Muh, MD, Principal Investigator — Henry Ford Health
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were assessed for eligibility and recruited for participation at their final preoperative clinic visit. Informed, written consent was obtained for eligible participants. Of 268 participants assessed for eligibility, 83 were included in the study. Of the 185 excluded participants, 69 declined participation while 116 met one of the exclusion criteria.
Pre-assignment Details: Included participants were not differentiated based on any factors before being randomized to a treatment group. Participant assignment to 1 of 2 treatment groups was performed using a computer generated random number sequence.
Units Other Than Participants: Shoulder
Groups:
- Non-opioid, Multimodal Protocol: Preoperatively, participants were treated with oral analgesics (400 mg celecoxib, 75 mg pregabalin, and 9 mg oxycodone extended-release). Intraoperatively, participants were administered 10 mg of dexamethasone and 1000 mg of acetaminophen intravenously in addition to a local periarticular injection (a solution containing 60 mg of 0.5% ropivacaine, 1 mg of epinephrine [1 mg/mL], and 30 mg of ketorolac). Postoperatively, all participants were discharged with oral medications that consisted of 4 mg dexamethasone twice daily for 4 days (participants that had an overnight hospital stay instead received a one-time 10 mg intravenously dexamethasone dose on postoperative day 1), 75 mg pregabalin twice daily for 14 days, 2 mg tizanidine every 6 hours for 14 days, 200 mg magnesium twice daily for 14 days, 600 mg ibuprofen every 6 hours (not to exceed 3200 mg per day) for 1 month, and 975 mg acetaminophen every 8 hours (not to exceed 3000 mg per day) for 1 month.
- Opioid Protocol: Preoperatively, participants were treated with oral analgesics (400 mg celecoxib, 75 mg pregabalin, and 9 mg oxycodone extended-release). Intraoperatively, participants were administered 10 mg of dexamethasone and 1000 mg of acetaminophen intravenously in addition to a local periarticular injection (a solution containing 60 mg of 0.5% ropivacaine, 1 mg of epinephrine [1 mg/mL], and 30 mg of ketorolac). Postoperatively, participants were discharged with oral medications that consisted of 4 mg dexamethasone twice daily for 4 days (participants that had an overnight hospital stay instead received a one-time 10 mg intravenously dexamethasone dose on postoperative day 1), 75 mg pregabalin twice daily for 14 days, 2 mg tizanidine every 6 hours for 14 days, 200 mg magnesium twice daily for 14 days, 600 mg ibuprofen every 6 hours (not to exceed 3200 mg per day) for 1 month, and 975 mg acetaminophen every 8 hours (not to exceed 3000 mg per day) for 1 month. Participants were given an additional prescription for 28 pills of 5 mg oxycodone to be taken for severe pain (≥ 6 on visual analog scale [VAS]). Participants in this treatment group could opt for receiving a rescue opioid prescription of 28 pills of 5 mg oxycodone if they felt that their pain was not sufficiently managed (severe pain, ≥ 6 on VAS).
Period: Overall Study
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Started | 41; 41 Shoulder | 42; 42 Shoulder
Completed | 38; 38 Shoulder | 40; 40 Shoulder
Not Completed | 3; 3 Shoulder | 2; 2 Shoulder
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Population: loss to follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [66 to 73] | 69 [65 to 72] | 70 [65 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 20 | 22 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31 | 33 | 64
  Black | 7 | 5 | 12
  Hispanic | 0 | 1 | 1
  Other | 0 | 1 | 1
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.9 [26.7 to 33.4] | 29.1 [26.6 to 33.6] | 29.9 [27.2 to 33.0]
Procedure Type [Count of Participants; unit: Participants] — Type of surgery, anatomic total shoulder arthroplasty (TSA) vs reverse total shoulder arthroplasty (RTSA)
  Participants
    TSA | 2 | 6 | 8
    RTSA | 35 | 34 | 69
tobacco use [Count of Participants; unit: Participants]
  Never | 26 | 25 | 51
  Former | 11 | 13 | 24
  Current | 1 | 2 | 3
Diabetes status [Count of Participants; unit: Participants]
  Yes | 8 | 9 | 17
  No | 30 | 31 | 61
Insulin dependence status [Count of Participants; unit: Participants]
  Yes | 3 | 5 | 8
  no | 35 | 35 | 70
hypertension [Count of Participants; unit: Participants]
  yes | 26 | 25 | 51
  no | 12 | 15 | 27
chronic kidney disease [Count of Participants; unit: Participants]
  yes | 2 | 1 | 3
  no | 36 | 39 | 75
Worker's compensation [Count of Participants; unit: Participants] — Is the patient paying for the surgery with a worker's compensation claim?
  Participants
    Yes | 1 | 0 | 1
    No | 37 | 40 | 77

OUTCOME MEASURES:

1. Primary Outcome: Pain Levels
Description: Patients record pain levels using a Visual analog scale for 10 days post-operatively. On each day, patients report their pain level via an automated text messaging service in the morning, afternoon, and the evening. A mean pain level is calculated from all scores reported by a patient in the first 10 days postoperatively. Patients will use a 0-10 scale along with visuals to indicate their level of pain with 0 being no pain at all and 10 being the worst pain possible. Lower scores indicate better outcomes.
Time Frame: The first 10 days postoperatively
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: score
Units Other Than Participants: shoulders
Groups:
- Non Opioid, Multimodal Protocol: Preoperatively, participants were treated with oral analgesics (400 mg celecoxib, 75 mg pregabalin, and 9 mg oxycodone extended-release). Intraoperatively, participants were administered 10 mg of dexamethasone and 1000 mg of acetaminophen intravenously in addition to a local periarticular injection (a solution containing 60 mg of 0.5% ropivacaine, 1 mg of epinephrine [1 mg/mL], and 30 mg of ketorolac). Postoperatively, all participants were discharged with oral medications that consisted of 4 mg dexamethasone twice daily for 4 days (participants that had an overnight hospital stay instead received a one-time 10 mg intravenously dexamethasone dose on postoperative day 1), 75 mg pregabalin twice daily for 14 days, 2 mg tizanidine every 6 hours for 14 days, 200 mg magnesium twice daily for 14 days, 600 mg ibuprofen every 6 hours (not to exceed 3200 mg per day) for 1 month, and 975 mg acetaminophen every 8 hours (not to exceed 3000 mg per day) for 1 month.
Arm/Group | Non Opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
score | 2.4 (1.7) | 2.3 (1.6)
Statistical Analysis 1: Comparison: Non Opioid, Multimodal Protocol vs Opioid Protocol; Test type: Equivalence — Mean scores between the two treatment groups will be compared using the Mann Whitney U test; p = 0.52, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.52

2. Secondary Outcome: Patient-Reported Outcomes Scores (PROMs) for Upper Extremity Pain Interference
Description: Patient-Reported Outcome Measures (PROMs) scores for upper extremity pain and how it interferes with the patients daily life. A T-score is given with a standard deviation based on the patients answers to the computerized adaptive test. The metrics have been designed to conform to a 10 - 90-point scale, with a score of 50 representing the mean of the population at large, 10 representing the minimum, and 90 representing the maximum function. A higher T-score represents higher pain interference (worse outcomes). Patient-Reported Outcomes Measurement Information System Physical Interference (PROMIS-PI) once every night for 10 days post-operatively.
Time Frame: Preoperatively, 10 days postoperatively, 6 weeks postoperatively, and 3 months postoperatively
Population: Loss to follow-up; participant did not fill out questionnaire
Measure: Mean (Standard Deviation); unit: T-score
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
T-score
  Preoperative | 62.4 (5.3) | 60.9 (4.6)
  10 days postoperative: number analyzed (Participants) | 32 | 36
  10 days postoperative: number analyzed (shoulders) | 32 | 36
  10 days postoperative | 60.9 (7.3) | 60.27 (6.5)
  6 weeks postoperatively: number analyzed (Participants) | 36 | 40
  6 weeks postoperatively: number analyzed (shoulders) | 36 | 40
  6 weeks postoperatively | 58.7 (7.6) | 55.7 (7.5)
  3 months postoperatively: number analyzed (Participants) | 34 | 35
  3 months postoperatively: number analyzed (shoulders) | 34 | 35
  3 months postoperatively | 51 (8.4) | 52.7 (8.3)

3. Secondary Outcome: Patient-Reported Outcomes Scores (PROMs) for Upper Extremity Function
Description: Patient-Reported Outcome Measures (PROMs) scores for upper extremity function. A T-score is given with a standard deviation based on the patients answers to the computerized adaptive test. The metrics have been designed to conform to a 0 - 100-point scale, with a score of 50 representing the mean of the population at large, 0 representing the minimum, and 100 representing the maximum function.
Time Frame: Preoperatively, 6 weeks postoperatively, and 3 months postoperatively
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: T-score
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
T-score
  preoperative | 30.2 (5.8) | 32.6 (5.7)
  6 weeks postoperative: number analyzed (Participants) | 35 | 40
  6 weeks postoperative: number analyzed (shoulders) | 35 | 40
  6 weeks postoperative | 33.5 (6.7) | 32.5 (6)
  3 months postoperative: number analyzed (Participants) | 32 | 34
  3 months postoperative: number analyzed (shoulders) | 32 | 34
  3 months postoperative | 39 (8.6) | 37 (8.5)

4. Secondary Outcome: Patient-Reported Outcomes Scores (PROMs) for Depression
Description: Patient-Reported Outcome Measures (PROMs) scores for depression. A T-score is given with a standard deviation based on the patients answers to the computerized adaptive test. The metrics have been designed to conform to a 10 - 90-point scale, with a score of 50 representing the mean of the population at large, 10 representing the minimum, and 90 representing the maximum function. A higher T-score represents higher increased depression (worse).
Time Frame: Preoperatively, 6 weeks postoperatively, and 3 months postoperatively
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: T-score
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
T-score
  preoperative | 47.9 (10.2) | 46 (7.8)
  6 weeks postoperative: number analyzed (Participants) | 33 | 36
  6 weeks postoperative: number analyzed (shoulders) | 33 | 36
  6 weeks postoperative | 43.2 (9.5) | 44.4 (9.5)
  3 months postoperative: number analyzed (Participants) | 32 | 33
  3 months postoperative: number analyzed (shoulders) | 32 | 33
  3 months postoperative | 42.2 (8.3) | 45.5 (7.7)

5. Secondary Outcome: American Shoulder and Elbow Score
Description: This is a patient reported outcome measure meant to assess participant shoulder function and pain. The score ranges from 0 to 100, with 0 representing a combination of poor shoulder function and high pain burden and 100 representing a lack of shoulder pain or functional deficit. The score is obtained by combining two subscale scores which are weighted equally. The first subscale is the visual analog scale, which asks participants to rate their pain on a scale of 0 to 10. A score of 0 indicates no pain and a score of 10 indicates the worst pain imaginable. The second subscale is the activities of daily living questionnaire. This questionnaire is composed of 10 questions, each asking about a specific activity of daily living related to shoulder function. For each question, the answer choices include: unable to do (0 points); very difficult to do (1 point); somewhat difficult (2 points); not difficult (3 points).
Time Frame: Preoperatively, 6 weeks postoperatively, and 3 months postoperatively
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
Scores on a scale
  Preoperative: number analyzed (Participants) | 36 | 36
  Preoperative: number analyzed (shoulders) | 36 | 36
  Preoperative | 43.9 (16.6) | 47.5 (20)
  6 weeks postoperative: number analyzed (Participants) | 33 | 32
  6 weeks postoperative: number analyzed (shoulders) | 33 | 32
  6 weeks postoperative | 64 (17.6) | 65.2 (18.9)
  3 months postoperative: number analyzed (Participants) | 19 | 27
  3 months postoperative: number analyzed (shoulders) | 19 | 27
  3 months postoperative | 71.1 (20.3) | 75 (16.5)

6. Primary Outcome: Morphine Milligram Equivalents
Description: The morphine milligram equivalents (MMEs) of opioids consumed will be recorded.
Time Frame: The first 10 days postoperatively.
Population: loss to follow-up
Measure: Mean (Standard Deviation); unit: morphine milligram equivalent
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
morphine milligram equivalent | 0.4 (1.35) | 3.7 (5.07)
Statistical Analysis 1: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Test type: Equivalence — Mean scores will be compared between the groups using the Mann Whitney U test; p < 0.001, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.001

7. Secondary Outcome: Shoulder Arthroplasty Smart Score (SAS)
Description: This is a score from 0 to 100 meant to represent the level of participant shoulder function. 0 represents the most poor function, and 100 the best possible score for function. The score is determined by combining three range of motion measures and 3 questions which are answered on a scale of 0 to 10. The three range of motion measures include forward flexion, internal rotation, and external rotation. The remaining three questions are as follows: What is your average pain on a daily basis?; What is your ability to use your affected shoulder on a daily basis?; What is your average pain when lying on affected side?
Time Frame: preoperatively; 6 weeks postoperatively; 3 months postoperatively
Population: Loss to follow-up
Measure: Mean (Standard Deviation); unit: Score
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
Score
  preoperative: number analyzed (Participants) | 32 | 33
  preoperative: number analyzed (shoulders) | 32 | 33
  preoperative | 44 (14.3) | 51.5 (10)
  6 weeks postoperative: number analyzed (Participants) | 13 | 16
  6 weeks postoperative: number analyzed (shoulders) | 13 | 16
  6 weeks postoperative | 58 (7.7) | 60.7 (12.4)
  3 months postoperative: number analyzed (Participants) | 22 | 25
  3 months postoperative: number analyzed (shoulders) | 22 | 25
  3 months postoperative | 70.1 (9.8) | 67.3 (10.3)

8. Secondary Outcome: Medication Side Effects
Description: The side effects were assessed to see whether they were present or not in the first 10 days postoperatively. They include constipation, nausea, diarrhea, upset stomach drowsiness, and loopiness
Time Frame: First 10 days postoperatively
Population: loss to follow-up
Measure: Mean (Standard Deviation); unit: days affected
Units Other Than Participants: shoulders
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
Number analyzed (shoulders) | 38 | 40
days affected
  constipation | 1.4 (2) | 2.3 (2.2)
  nausea | 0.5 (1) | 0.3 (0.6)
  diarrhea | 0.2 (0.8) | 0.1 (0.3)
  upset stomach | 0.8 (1.7) | 0.9 (1.7)
  drowsiness | 1.4 (2) | 2.3 (2.2)
  loopiness | 2 (2.8) | 2.5 (2.9)
Statistical Analysis 1: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Comparing the distribution of the number of days participants were affected by each side effect; Test type: Equivalence — mann-whitney U; p = 0.06, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.06
Statistical Analysis 2: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Comparing the distribution of the number of days participants were affected by each side effect; Test type: Equivalence — mann-whitney U; p = 0.73, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.73
Statistical Analysis 3: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Comparing the distribution of the number of days participants were affected by each side effect; Test type: Equivalence — mann-whitney; p = 0.61, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.61
Statistical Analysis 4: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Comparing the distribution of the number of days participants were affected by each side effect; Test type: Equivalence — mann-whitney; p = 0.47, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.47
Statistical Analysis 5: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Comparing the distribution of the number of days participants were affected by each side effect; Test type: Equivalence — mann-whitney; p = 0.47, Wilcoxon (Mann-Whitney); mann-whitney = 0.47
Statistical Analysis 6: Comparison: Non-opioid, Multimodal Protocol vs Opioid Protocol; Comparing the distribution of the number of days participants were affected by each side effect; Test type: Equivalence — mann-whitney; p = 0.74, Wilcoxon (Mann-Whitney); Mann-Whitney = 0.74

9. Secondary Outcome: Number of Patients Who Required Reoperation
Description: Whether or not patients required another operation.
Time Frame: To 2 years postoperative
Population: loss to follow-up
Measure: Number; unit: participants
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
Number analyzed (Participants) | 38 | 40
participants | 0 | 1

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to two years postoperatively
Arm/Group | Non-opioid, Multimodal Protocol | Opioid Protocol
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 2/38 | 2/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-opioid, Multimodal Protocol (N=38) | Opioid Protocol (N=40)
acromion fracture (Musculoskeletal and connective tissue disorders) | 2 | 2 — Event is a complication of shoulder arthroplasty

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/47/NCT05488847/Prot_SAP_ICF_000.pdf